CLINICAL TRIAL: NCT07123792
Title: Comparison of Different Intracanal Medicaments on Post-operative Pain in Teeth With Symptomatic Apical Periodontitis: A Randomised Controlled Trial
Brief Title: Effect of Intracanal Medicaments on Post-Operative Pain in Symptomatic Apical Periodontitis: An RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, fatimaharshad, Principal investigator, College of Physicians and Surgeons Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dr Fatimah
Record Dates: First submitted 2025-07-31; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Calcium Hydroxide; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Calcium Hydroxide group (Experimental): Participants in this group will receive 20% calcium hydroxide paste as the intracanal medicament after root canal instrumentation. The medicament will be placed using a Lentulo spiral, excess removed from the chamber, and the tooth sealed with glass ionomer cement. Pain will be assessed at 0, 6, 24, and 48 hours postoperatively.
  Interventions: Drug: Calcium Hydroxide (20%)
- Chlorhexidine group (Experimental): Participants in this group will receive 2% chlorhexidine gel as the intracanal medicament following canal preparation. It will be placed with a Lentulo spiral and sealed in the same manner. Postoperative pain will be evaluated at the same intervals.
  Interventions: Drug: Chlorhexidine Gel (2%)
- Modified triple antibiotic paste (Experimental): Participants in this group will receive a modified triple antibiotic paste made from ciprofloxacin, metronidazole, and clindamycin in a 1:1:1 ratio by weight. The paste will be placed inside the canal using a Lentulo spiral and sealed as per protocol. Pain will be recorded at 0, 6, 24, and 48 hours post-treatment.
  Interventions: Drug: Modified Triple Antibiotic Paste

INTERVENTIONS:
Drug: Calcium Hydroxide (20%) — A 20% calcium hydroxide paste will be placed as an intracanal medicament following root canal instrumentation. Applied using a Lentulo spiral, excess is removed, and the tooth is sealed with a glass ionomer temporary restoration.
  Other Names: Modified triple antibiotic paste
  Arms: Calcium Hydroxide group
Drug: Chlorhexidine Gel (2%) — A 2% chlorhexidine gel will be used as an intracanal medicament following canal preparation. It will be delivered with a Lentulo spiral, cleaned from the chamber, and the tooth sealed.
  Other Names: Calcium hyroxide
  Arms: Chlorhexidine group
Drug: Modified Triple Antibiotic Paste — A modified triple antibiotic paste consisting of ciprofloxacin, metronidazole, and clindamycin (1:1:1 by weight) will be placed in the canal using a Lentulo spiral. The excess paste will be removed, and the cavity will be sealed with temporary restorative material.
  Other Names: Chlorhexidine
  Arms: Modified triple antibiotic paste

SUMMARY:
Comparison of different intracanal medicaments during root canal treatment to assess their effect on post-operative pain in teeth with Symptomatic Apical Periodontitis

DETAILED DESCRIPTION:
Pain is the most common clinical symptom associated with endodontic treatment. Symptomatic apical periodontitis (SAP) results in significant post-operative discomfort due to microbial invasion and inflammatory changes in periapical tissues. Intracanal medicaments are used to reduce microbial load and inflammation between treatment appointments, potentially reducing post-treatment pain. This study investigates the comparative effectiveness of three commonly used intracanal medicaments in reducing pain following biomechanical preparation:

Group 1: Calcium hydroxide (CH)

Group 2: Chlorhexidine gel (CHX 2%)

Group 3: Modified Triple Antibiotic Paste (TAP) - a combination of ciprofloxacin, clindamycin, and metronidazole in 1:1:1 ratio

A total of 480 participants with single-rooted teeth diagnosed with symptomatic apical periodontitis will be randomly assigned into three groups (160 in each group). Endodontic treatment will be performed by a single operator under standard protocols. No systemic analgesics or antibiotics will be prescribed. Pain assessment will be done using the Wong-Baker FACES Pain Rating Scale (0-10), and recorded at baseline (0 h), 6 h, 24 h, and 48 h after treatment.

The study aims to provide evidence on the most effective intracanal medicament to minimize post-operative pain, improving patient outcomes and guiding clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Single rooted teeth (Anterior or posterior)
* Teeth with acute symptomatic apical periodontitis

Exclusion Criteria:

* Non-restorable teeth, presence of endo-perio lesions, teeth with acute or chronic apical abcess, teeth with internal/external root resorption
* Teeth with anatomical difficulties like open apices, calcified canals, dilacerations
* Patients with parafunctional habits
* Patients who were allergic to medications that were used in the study
* Patients who were taking medicines that could influence pain perception
* Patients that had any serious medical illness or with systemic disorders

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 480 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-05-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Post-operative Pain Intensity Measured Using the Wong-Baker FACES Pain Rating Scale (WFPRS) | At baseline (0 hours), 6 hours, 24 hours, and 48 hours post-operatively
  Pain intensity will be assessed using the Wong-Baker FACES Pain Rating Scale (WFPRS), a validated 6-point facial expression scale. The scale ranges from 0 (no pain) to 10 (worst pain), with corresponding facial images used to help patients subjectively rate their pain. This tool will be used during follow-up calls to determine the patient's level of pain after root canal instrumentation and medicament placement.
  Units of Measurement:
  Score range: 0-10 (intervals of 2)

CONTACTS AND LOCATIONS:
Overall Officials: Beenish Qureshi, BDS, FCPS, Study Chair — HITEC-Institute of Medical Sciences
Locations (1):
- Dental hospial, Hitec-IMS, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan AM, Gangoo IKA, Ali NA, Khan M, Javed MQ, AlAttas MH, Abulhamael AM, Bahammam HA, Alsofi L, Yahya RSA. The Effect of Calcium Hydroxide, Triple Antibiotic Paste and Chlorhexidine on Pain in Teeth with Symptomatic Apical Periodontitis: A Randomised Controlled Trial. Int J Environ Res Public Health. 2023 Feb 10;20(4):3091. doi: 10.3390/ijerph20043091. PMID 36833788